CLINICAL TRIAL: NCT05375825
Title: Phase I Evaluation of Immunotoxin LMB-100 Administered by Normothermic, Intrapleural Perfusion Following Cytoreductive Surgery in Participants With Pleural Mesotheliomas, or Pleural Effusions From Cancers Expressing Mesothelin
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000062; 000062-C
Record Dates: First submitted 2022-05-14; First posted 2022-05-17 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Malignant Pleural Mesotheliomas (Mpm); Malignant Pleural Effusions (Mpe); Epithelial Tumors, Malignant; Pleural Effusions, Malignant; Mesothelin (Msln)
Keywords: Pleural Metastases; Malignant Pleural Mesotheliomas (Mpm); Malignant Pleural Effusions (Mpe); Anti-Mesothelin; Mesothelin-Positive Malignancy; Progression Free Survival (Pfs); Overall Survival (Os)
MeSH Terms: conditions — Mesothelioma, Malignant; Pleural Effusion, Malignant; Myeloproliferative Disorder, Chronic, with Eosinophilia; Carcinoma | interventions — Cytoreduction Surgical Procedures; LMB-100

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Dose Escalation (Experimental): LMB-100 at escalating/de-escalating doses + MSLN testing
  Interventions: Procedure: Cytoreductive surgery; Drug: LMB-100; Diagnostic Test: Immunohistochemical Assay for Mesothelin
- 2/ Dose Expansion (Experimental): LMB-100 at the MTD + MSLN testing
  Interventions: Procedure: Cytoreductive surgery; Drug: LMB-100; Diagnostic Test: Immunohistochemical Assay for Mesothelin

INTERVENTIONS:
Procedure: Cytoreductive surgery — Cytoreductive surgery: minimally invasive (VATS/robotic) or open (thoracotomy)
Drug: LMB-100 — 1000 mcg/mL (DL1) post-operative dose as a single 90-minute normothermic intrathoracic perfusion using a closed circuit and roller pump with a heat exchanger following maximal cytoreductive surgery
Diagnostic Test: Immunohistochemical Assay for Mesothelin — Performed at screening to determine mesothelin expression; separate testing of tumor mesothelin expression will be assessed retrospectively in resected tumor tissues. The device is not diagnostic; protocol assessment of mesothelin expression status will only be used to help to increase the possibility that all persons enrolling on the study might derive benefit from therapy.

SUMMARY:
Background:

Cancers that spread into the thin tissue lining your lungs (pleura) cause serious illness. They often recur when removed. These tumors include malignant pleural mesothelioma (MPM), caused by exposure to asbestos and related fibers. Malignant pleural effusions (MPEs) are caused when cancers in other parts of the body spread to the lungs and pleura. Many people diagnosed with pleural tumors survive less than a year.

Objective:

To test the safety of a study drug (LMB-100) in people. LMB-100 may help stop pleural tumors from recurring after surgery.

Eligibility:

People aged 18 years or older diagnosed with MPM or related cancer that has spread into the pleura.

Design:

Participants will undergo screening. They will have a physical exam with blood and urine tests. They will have CT scans. They will have tests that measure the how their heart and lungs function. They will provide a sample of tumor tissue to determine if their tumor expresses a protein called mesothelin.

Participants will undergo standard surgery to maximally remove the plural tumors. Then they will have LMB-100 pumped into their chest. The liquid will rinse the chest wall, diaphragm, heart sac, and surface of the lungs for 90 minutes. Then the liquid will be drained and the surgical incisions closed. The participants will be under anesthesia during this procedure.

Participants will remain in the intensive care unit for a least 48 hours. They will remain in the hospital for up to a week or more until recovered enough to be safely discharged.

Participants will return for regular follow-up visits for 2 years.

DETAILED DESCRIPTION:
Background

* Malignant pleural mesotheliomas (MPM) are aggressive cancers with a high predilection for intrapleural recurrences despite potentially curative resections.
* Pleural metastases and associated malignant pleural effusions (MPE) cause considerable morbidity and mortality in patients with lung and esophageal cancers, gastrointestinal, pancreatic, and ovarian carcinomas, as well as sarcomas.
* Mesothelin (MSLN), a tumor differentiatio antigen, is expressed in over 95% of epithelioid MPM, as well as 80% of thymic carcinomas, 50% of lung and gastroesophageal cancers, 75% of pancreatic carcinomas, and 30% of ovarian carcinomas and synovial sarcomas.
* Mesothelin is an attractive target for cancer therapy due to its limited expression in normal human tissues and effects on invasion and metastasis of cancer cells.
* LMB-100 is a novel recombinant anti-mesothelin immunotoxin containing a humanized fragment of an anti-mesothelin Fab conjugated to a de-immunized Pseudomonas exotoxin A (PEA) which exhibits broad activity against cancer lines and tumor xenografts expressing mesothelin.
* Despite de-immunizing modifications, LMB-100 still induces neutralizing antibodies that prevent repeated systemic administration of this immunotoxin.
* Local (intraperitoneal) administration of LMB-100 can eradicate low-volume carcinomatosis in a murine model of minimal residual disease.
* Conceivably, intracavitary administration of LMB-100 following cytoreductive surgery may enhance local control of pleural-based malignancies that express mesothelin while minimizing systemic exposure of the immunotoxin.

Primary Objective

-To identify maximum tolerated dose (MTD) and evaluate the toxicities of LMB-100 administered by 90-minute normothermic, intrapleural perfusion in participants with mesothelin-positive MPM, or MPE from cancers that express mesothelin.

Eligibility

* Age >= 18 years
* Histologically confirmed mesothelioma, or other mesothelin-positive malignancy metastatic to the pleura, potentially amenable to cytoreductive surgery and subsequent intrapleural perfusion.
* No systemic or local therapy for their malignancy within 3 weeks prior to protocol treatment.
* Adequate organ function and cardiopulmonary reserve to tolerate intended resection.
* No active infections.
* No active central nervous system (CNS) metastases.

Design

* Participant s will undergo maximal cytoreductive surgery for their malignancies by open or minimally invasive procedures as dictated by histologic, anatomic, and physiologic parameters.
* Thereafter, LMB-100 will be administered by 90-minute normothermic intrathoracic perfusion using a closed circuit and roller pump with a heat exchanger.
* LMB-100 levels will be measured in pulmonary lavage and plasma.
* The dose of LMB-100 will be increased using a 3 plus 3 design to define MTD.
* Once the MTD has been defined, the enrollment will be expanded to more fully define toxicities and evaluate time to disease progression and overall survival (OS) using 2 separate cohorts of participants with MPM and pleural effusions from other malignances (MPE).
* The accrual ceiling will be set at 42.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Histologically confirmed by the Laboratory of Pathology (LP), CCR, NCI mesothelinpositive malignancy arising from or metastatic to the pleura that is potentially amenable to cytoreductive surgery (R0-R2) and subsequent intrapleural perfusion based on standard of care (SOC) imaging.
2. Participants with biphasic MPM must have a < 50% sarcomatoid component.
3. Participants with MPE from extra-thoracic disease may be eligible provided these sites are controlled and are less threatening than the pleural involvement LENT score >=2 .
4. Participants with stage IV cancers affecting the pleura with MPE must have received firstline standard of care systemic treatment for their malignancies.
5. MPM participants must not have received any local or systemic therapy for their disease.
6. All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure must have resolved to Grade <= 1 except hemoglobin (Hgb) <= Grade 2, alopecia (any grade), and <= Grade 2 peripheral neuropathy.
7. Age >18 years.
8. ECOG performance status of < 2.
9. Participants must have adequate pulmonary reserve evidenced by post-operative predicted FEV1 and adjusted DLCO >= 40% predicted.
10. Room air oxygen saturation >= 90%; otherwise pCO2 <= 45 and pO2 >= 60 on room air arterial blood gas (ABG).
11. Adequate organ and marrow function as defined below:

    * leukocytes >= 3,000/mcL
    * absolute neutrophil count >= 1,500/mcL (without transfusion or cytokine support)
    * absolute lymphocyte count > 800/mcL
    * platelets >= 100,000/mcL
    * Hgb >= 9 g/ dL (with transfusion if necessary, within 1 week prior to treatment)
    * serum albumin >= 2.0 mg/dL
    * AST/ALT <= 2.5 X institutional ULN
    * creatinine clearance (eGFR) >= 50 mL/min/1.73 m^2 by Cockcroft-Gault formula
    * INR <= 1.5 x ULN
    * TSH, T3 and T4 within normal limits (WNL) per institutional criteria
    * random serum cortisol within normal limits (WNL) per institutional criteria
    * total bilirubin < 1.5 X institutional ULN (excluding Gilbert s Syndrome)
12. No active brain metastases. Participants with a history of brain metastases except those with meningeal carcinomatosis or leptomeningeal disease may be eligible for treatment a minimum of 1 week following completion of gamma knife or whole-brain radiotherapy, or 4 weeks

    following surgical resection of brain metastases provided post-treatment MRI scan reveals no evidence of active disease and no ongoing need for systemic steroids.
13. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) at the study entry, for the duration of study treatment and up to 4 months (women) or 2 months (men) after the last dose of the study drug.
14. Breastfeeding participants must be willing to discontinue breastfeeding from study enrollment through two months after the LMB-100 perfusion.
15. HBV-infected participants must be on antivirals and have HBV DNA <100 IU/mL. HCV-infected participants can be enrolled if HCV RNA level is undetectable.
16. The ability of the participant to understand and the willingness to sign a written informed consent.
17. Participants must be enrolled into protocol 06C0014 "Prospective Evaluation of Genetic and Epigenetic Alterations in Patients with Thoracic Malignancies".
18. Participants must provide acceptable archival tumor samples or have at least 1 focus of disease that is amenable to tumor biopsy if necessary for confirmation of histology, and assessment of mesothelin expression.

EXCLUSION CRITERIA:

1. Active smokers.
2. Participants receiving systemic steroids other than physiologic replacement doses or inhaled corticosteroids (<= 20 mg of dexamethasone a day [or equivalent]) for <= 7 consecutive days prior to treatment initiation).
3. Treatment with chemotherapy, targeted therapy, immunotherapy, radiation, or surgery to an index lesion within three weeks prior to commencing protocol therapy, excluding minor surgical procedures (i.e. VATS/thoracentesis/PleurX catheter placement to palliate

   MPE).
4. Treatment with another investigational agent within four weeks prior to commencing protocol therapy.
5. History of allergic reactions attributed to compounds of chemical or biologic composition similar to LMB-100 or SS1P including pseudomonas endotoxin.
6. Clinically significant cardiovascular/cerebrovascular disease as follows: cerebral vascular accident/stroke (within 6 months prior to treatment initiation) or myocardial infarction (within 6 months prior to treatment initiation) unless revascularized, unstable angina, congestive heart failure (New York Heart Association Classification Class >= II), serious cardiac arrhythmia, abnormal ejection fraction (echocardiogram [ECHO]) <= 40%, clinically significant bleeding or clinically significant pulmonary embolism.
7. History of pneumonitis (idiopathic or drug-induced) unless cleared by pulmonary consultants.
8. Receipt of any organ transplantation, including allogeneic stem-cell transplantation, except transplants that do not require immunosuppression (e.g., corneal transplant, hair transplant).
9. HIV-infected participants. Participants on stable doses of antiretroviral therapy whose HIV RNA is below level of quantification are eligible.
10. Active COVID-19 infection.
11. Active infections requiring systemic therapy.
12. An additional malignancy that is progressing or requires active treatment.
13. Pregnancy
14. Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Identify maximum tolerated dose (MTD) and evaluate the toxicities of LMB-100 administered by 90-minute normothermic, intrapleural perfusion in participants with mesothelin-positive MPM, or MPE from cancers that express mesothelin | 21 days
  List of adverse event frequency, type, and grade Safety data based on toxicity grades and types of toxicity will be reported by dose level during dose escalation.

SECONDARY OUTCOMES:
Determine 2 year progression free survival (PFS), and 3 year overall survival of participants following intrapleural LMB-100 perfusion | at initial perfusion, every 3 months (+/- 2 weeks), to time of documented clinical recurrence and/or death
  Cytoreductive surgery until time of documented clinical recurrence (radiographically or pathologically) Progression free survival (PFS): 2 year PFS probability will be calculated from the on-study date through 2 years after initiation of study therapy using the Kaplan-Meier method. Overall Survival (OS): 3 year OS probability from the on-study date through 3 years after initiation of study therapy
Identify pharmacokinetics of LMB-100 administered by 90-minute normothermic, intrapleural perfusion | Pre-dose, completion of perfusion, and 1, 3, 24 hours after start of perfusion
  Pharmacokinetic accumulation of free and total plasma concentrations of LMB-100 will be measured using validated ligand-binding assays analyzed in the blood (plasma)and pulmonary lavage at protocol time points. Analyses will be performed retrospectively in batched samples or at the end of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. @@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000062-C.html